CLINICAL TRIAL: NCT03008512
Title: A Phase II Study of Weekly Genexol-PM in Patients With Advanced Hepatocelluar Carcinoma After Failure of Sorafenib
Brief Title: A Phase II Study of Weekly Genexol-PM in Patients With Hepatocelluar Carcinoma After Failure of Sorafenib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Young Saing Kim, Assistant professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: weGePM-HCC
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Liver Neoplasms; Antineoplastic Agents; Carcinoma, Hepatocellular; Genexol-PM; Neoplasms by Site; Sorafenib; Liver Diseases; Digestive System Neoplasms
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms by Site; Liver Diseases; Digestive System Neoplasms | interventions — genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genexol-PM (Experimental): Genexol-PM 100 mg/m2 intravenously for 1 hour on days 1, 8, and 15 of a 28-day cycle up to 8 cycles. Patients will receive study treatment until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Genexol-PM

INTERVENTIONS:
Drug: Genexol-PM
  Other Names: Cremophor-free, polymeric micelle-formulated paclitaxel

SUMMARY:
This study evaluate activity and safety profile of weekly Genexol-PM in patients with advanced hepatocellular carcinoma for whom sorafenib treatment failed. Patients will receive Genexol-PM on days 1, 8, and 15 every 4 weeks.

DETAILED DESCRIPTION:
Hepatocelluar carcinoma (HCC) is a highly vascular neoplasm characterized by arterial enhancement on CT or MRI. Angiogenesis provides a target for novel prognostic and therapeutic approaches to HCC. Sorafenib is the standard 1st-line therapy shown to significantly improve overall survival in advanced HCC. However, sorafenib benefits are mostly transient and modest. In addition, sorafenib is associated with major toxicities, and about 30% of patients stop it because of intolerance. Effective therapies are needed for patients who experience progression during or after receiving sorafenib or who have sorafenib intolerance. Paclitaxel has an antiagiogenic activity and weekly administration of paclitaxel is considered to have enhanced efficacy over 3-weekly administration due to greater drug exposure or a direct antiangiogenic effect. A previous phase I study showed that weekly paclitaxel has activity in hepatocellular carcinoma and further investigation in phase II trials is warranted. Genexol-PM, a cremophor-free, polymeric micelle-formulated paclitaxel, is believed to be superior to conventional paclitaxel in terms of the obviation of premedication and the delivery of higher paclitaxel doses without additional toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of hepatocellular carcinoma (HCC) based on either

   1. histopathologic or cytologic findings
   2. a diagnosis of cirrhosis and HCC with classical imaging characteristics (at least a 3-phase liver protocol CT or MRI and a lesion that demonstrates arterial enhancement and washes out in the venous phase)
2. Previous sorafenib treatment for at least 14 days and discontinuation of sorafenib treatment prior to inclusion
3. Radiologic confirmation of disease progression during or after discontinuation of sorafenib treatment or discontinuation of sorafenib due to intolerance despite appropriate supportive care
4. Barcelona Clinic Liver Cancer (BCLC) stage C or BCLC stage B disease not amenable to locoregional therapy or refractory to locoregional therapy
5. ≥ 1 measurable lesion according to RECIST Version 1.1
6. ≥ 20 year of age
7. ECOG performance status ≤ 2
8. Child-Pugh score ≤ 7
9. Informed consent prior to study
10. Adequate organ function

    1. Hepatic: bilirubin ≤ 1.5 times upper limit of institutional normal value (ULN), AST or ALT ≤ 5 x ULN
    2. Renal: estimated creatinine clearance ≥ 60 mL/min
    3. Hematologic: hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1,500/μL, platelets ≥ 75,000/μL (In case of thrombocytopenia associated with hypersplenism in chronic liver disease, platelets ≥ 50,000/μL is allowed for participation at the physician's discretion.)
    4. Coagulation: prothrombin time (INR) ≤ 1.5, partial thrombin time (PTT) ≤ 5 seconds above the ULN

Exclusion Criteria:

1. Previous systemic chemotherapy for advanced disease (except previous biologic agents including VEGF inhibitors, TGF-beta inhibitors, or PD-1/PD-L1 blockers)
2. A history o f or current hepatic encephalopathy or clinically meaningful ascites
3. Grade 2 or more peripheral neuropathy
4. Prior liver transplant
5. History of any other cancer within 2 years (Patients with carcinoma in situ of any origin and patients with prior malignancy who are in remission and whose likelihood of recurrence is very low, may be eligible.)
6. A history of treatment with taxanes (paclitaxel or docetaxel)
7. Females who are pregnant or lactating
8. A know allergy or hypersensitivity reaction to any of the treatment components
9. Serious preexisting medical conditions that cannot adequately controlled with appropriate therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | Baseline to Objective Progression or Death from Any Cause (Approximately 12 Months)

SECONDARY OUTCOMES:
Progression-free survival | Baseline to Objective Progression or Death from Any Cause (Approximately 12 Months)
Overall survival | Baseline to Death from Any Cause (Approximately 12 Months)
Objective response rate | Baseline to Objective Progression (Approximately 12 Months)
Adverse events | Cycle 1 through Follow Up (Approximately 12 Months)
  NCI-CTCAE V4.03

CONTACTS AND LOCATIONS:
Overall Officials: Dong Bok Shin, Professor, Principal Investigator — Gachon University Gil Medical Center
Locations (2):
- South Korea (2):
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim TY, Kim DW, Chung JY, Shin SG, Kim SC, Heo DS, Kim NK, Bang YJ. Phase I and pharmacokinetic study of Genexol-PM, a cremophor-free, polymeric micelle-formulated paclitaxel, in patients with advanced malignancies. Clin Cancer Res. 2004 Jun 1;10(11):3708-16. doi: 10.1158/1078-0432.CCR-03-0655. PMID 15173077
- [Background] Strumberg D, Erhard J, Harstrick A, Klaassen U, Muller C, Eberhardt W, Wilke H, Seeber S. Phase I study of a weekly 1 h infusion of paclitaxel in patients with unresectable hepatocellular carcinoma. Eur J Cancer. 1998 Jul;34(8):1290-2. doi: 10.1016/s0959-8049(98)00054-9. PMID 9849493
- [Background] Bocci G, Di Paolo A, Danesi R. The pharmacological bases of the antiangiogenic activity of paclitaxel. Angiogenesis. 2013 Jul;16(3):481-92. doi: 10.1007/s10456-013-9334-0. Epub 2013 Feb 7. PMID 23389639
- [Background] Baird RD, Tan DS, Kaye SB. Weekly paclitaxel in the treatment of recurrent ovarian cancer. Nat Rev Clin Oncol. 2010 Oct;7(10):575-82. doi: 10.1038/nrclinonc.2010.120. Epub 2010 Aug 3. PMID 20683437